CLINICAL TRIAL: NCT02071797
Title: Early Targeted Brain Cooling in the Cath Lab Following Cardiac Arrest. Randomised Controlled Trial of RhinoChill Versus Blanketrol Intra-Hospital Induction of Therapeutic Hypothermia After Cardiac Arrest
Brief Title: Early Targeted Brain Cooling in the Cath Lab Following Cardiac Arrest
Acronym: COOLCATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B626; 12/EE/0472 (Other: REC)
Record Dates: First submitted 2014-01-27; First posted 2014-02-26 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Arrest
Keywords: Therapeutic Hypothermia; Cardiac Arrest; Randomised Controlled trial; Pilot study
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Blanketroll lll (Active Comparator): Cutaneous Cooling Blanket, Blanketroll lll, applied to cool patient to 32C. Standard care
  Interventions: Device: Induced Therapeutic Hypothermia
- Arm B - RhinoChill (Active Comparator): Intra nasal cooling system, RhinoChill, to cool patient to 32C - Standard care
  Interventions: Device: Induced Therapeutic Hypothermia

INTERVENTIONS:
Device: Induced Therapeutic Hypothermia — Head to head, direct comparator of two standard care devices/treatments (RhinoChill versus Blanketroll lll) to assess time to induced therapeutic hypothermia
  Other Names: RhinoChill will be compared with Blanketroll lll

SUMMARY:
The objective of the COOLCATH study is to compare the effect of the RhinoChill transnasal cooling system to current standard Blanketrol III cooling blanket in its ability to achieve therapeutic hypothermia (TH) induction for patients undergoing TH after cardiac arrest.

The COOLCATH study will be a prospective, open-label randomized controlled trial comparing induction of TH efficacy and outcomes of patients following cardiac arrest. Any patient with return of spontaneous circulation (ROSC) following a cardiac arrest within the Essex Cardiothoracic Centre (CTC), or who is brought to the Essex CTC and is a candidate for TH will be considered for this study.

DETAILED DESCRIPTION:
According to standard practice patients will be fully anaesthetised, intubated and ventilated. Patients will have a baseline tympanic temperature measurement taken and then will be randomized to receive induction of TH by either RhinoChill Transnasal cooling system, or standard care using the Blanketrol III cooling blanket.

All patients will have tympanic and oesophageal temperature measurement every 10 minutes until they reach TH (<34 degrees centigrade). Once TH is achieved, the RhinoChill will be discontinued, and all patients will then receive the Blanketrol III cooling blanket for maintenance of TH for the standard 24 hour period. If a patient achieves a core body temp of 34 degrees centigrade while undergoing RhinoChill cooling and is still on the cath lab table, the device will be turned to low flow to ensure that the temperature is maintained until a transfer to the Blanketrol system is possible. For patients that arrive in the ICU on RhinoChill with a temperature >34 (i.e. have not reached TH), these patients will have RhinoChill and blanket therapy until they reach <34 degrees centigrade when the RhinoChill will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Post cardiac arrest with Return of Spontaneous Circulation
3. Receiving therapeutic hypothermia as part of post-cardiac arrest care

Exclusion Criteria:

1. Cardiac arrest caused by trauma, head injury, massive haemorrhage, drug overdose, cerebrovascular accident, drowning, electric shock or hanging
2. Already hypothermic
3. Nasal obstruction preventing the insertion of a nasal catheter
4. Do Not Attempt to Resuscitate (DNAR) orders
5. Known terminal illness (eg. malignancy in the end stages)
6. Known or obvious pregnancy
7. Known coagulation disorder (except those induced by medication eg. Thrombolytics)
8. Known O2- dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to reduce tympanic temperature to < 34C | Day 1

SECONDARY OUTCOMES:
In hospital and 30 day mortality | Day 30
Length of Intensive Care Unit stay | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: John R Davies, MBBS MRCP, Study Director — BTUH
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Islam S, Hampton-Till J, Watson N, Mannakkara NN, Hamarneh A, Webber T, Magee N, Abbey L, Jagathesan R, Kabir A, Sayer J, Robinson N, Aggarwal R, Clesham G, Kelly P, Gamma R, Tang K, Davies JR, Keeble TR. Early targeted brain COOLing in the cardiac CATHeterisation laboratory following cardiac arrest (COOLCATH). Resuscitation. 2015 Dec;97:61-7. doi: 10.1016/j.resuscitation.2015.09.386. Epub 2015 Sep 26. PMID 26410565